CLINICAL TRIAL: NCT04271527
Title: Non-inferiority Randomized Controlled Trial of Cognitive Fusion Targeted Biopsy Versus Software-based Fusion Targeted Biopsy
Brief Title: Non-inferiority Randomized Controlled Trial of Cognitive Targeted Biopsy Versus Software Targeted Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Zibo Central Hospital (Other Government); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Henan university of CM (Unknown); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Peking University First Hospital (Other); The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CSTB-2019-001
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; cognitive fusion targeted biopsy; software-based fusion targeted biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive targeted biopsy (Experimental): a cognitive fusion targeted biopsy combined with a systematic biopsy
  Interventions: Procedure: cognitive fusion targeted biopsy
- software targeted biopsy (Active Comparator): software-based fusion targeted biopsy combined with a systematic biopsy
  Interventions: Procedure: cognitive fusion targeted biopsy

INTERVENTIONS:
Procedure: cognitive fusion targeted biopsy — A cognitive fusion targeted biopsy

SUMMARY:
This is a randomized controlled and non-inferiority trial in comparison of the cognitive fusion targeted biopsy between the software-based fusion targeted biopsy in the detection rate of clinically significant cancer in men suspected to have a PCa.

DETAILED DESCRIPTION:
This trial is a prospective, multi-centre, randomized controlled, and non-inferiority study in which all men suspicious to have clinically significant prostate cancer. This study aims to determine whether the cognitive fusion targeted biopsy is non-inferior to software-based fusion targeted biopsy in the detection rate of clinically significant cancer in men suspected to have a PCa.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. PSA increase to 4-20 ng/ml and/or abnormal DRE;
3. Sign the informed consent

Exclusion Criteria:

1. Have acute or chronic prostatitis
2. Contraindications to prostate biopsy
3. Contraindications to MRI
4. Other reasons that not suitable for this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 626 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
The detection rate of clinically significant prostate cancer for targeted biopsy | 5-6 weeks after signing the consent
  The proportion of men with a Gleason score ≥3+4 in pathological assessment for targeted biopsy samples

SECONDARY OUTCOMES:
The detection rate of any prostate cancer for targeted biopsy | 5-6 weeks after signing the consent
  The proportion of men with a Gleason score ≥3+3 in pathological assessment for targeted biopsy samples
The detection rate of clinically significant prostate cancer for combined biopsy | 5-6 weeks after signing the consent
  The proportion of men with a Gleason score ≥3+4 in pathological assessment for combined biopsy samples
The detection rate of any prostate cancer for combined biopsy | 5-6 weeks after signing the consent
  The proportion of men with a Gleason score ≥3+3 in pathological assessment for combined biopsy samples
Prostate volume | 5-6 weeks after signing the consent
  To measure the prostate volume by ultrasound and MRI
The detection rate of clinically significant prostate cancer in suspicious lesion with maximum diameter <0.5cm | 5-6 weeks after signing the consent
  Proportion of separate suspicious lesion with maximum diameter <0.5cm, detected ISUP grade group>=2 cancers by targeted biopsy only.
The detection rate of clinically significant prostate cancer in suspicious lesion with maximum diameter range from 0.5 ~ 1.0 cm | 5-6 weeks after signing the consent
  Proportion of separate suspicious lesion with maximum diameter range from 0.5 ~ 1.0 cm, detected ISUP grade group>=2 cancers by targeted biopsy only.
The detection rate of clinically significant prostate cancer in suspicious lesion with maximum diameter >1.0 cm | 5-6 weeks after signing the consent
  Proportion of separate suspicious lesion with maximum diameter >1.0 cm, detected ISUP grade group>=2 cancers by targeted biopsy only.
The detection rate of clinically significant prostate cancer in suspicious lesion with PI-RADS 3 | 5-6 weeks after signing the consent
  Proportion of separate suspicious lesion with PI-RADS 3, detected ISUP grade group>=2 cancers by targeted biopsy only.
The detection rate of clinically significant prostate cancer in suspicious lesion with PI-RADS 4 | 5-6 weeks after signing the consent
  Proportion of separate suspicious lesion with PI-RADS 4, detected ISUP grade group>=2 cancers by targeted biopsy only.
The detection rate of clinically significant prostate cancer in suspicious lesion with PI-RADS 5 | 5-6 weeks after signing the consent
  Proportion of separate suspicious lesion with PI-RADS 5, detected ISUP grade group>=2 cancers by targeted biopsy only.

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wang, MD, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He B, Li R, Li D, Huang L, Wen X, Yang G, Wang H. Study protocol for a single-centre non-inferior randomised controlled trial on a novel three-dimensional matrix positioning-based cognitive fusion-targeted biopsy and software-based fusion-targeted biopsy for the detection rate of clinically significant prostate cancer in men without a prior biopsy. BMJ Open. 2021 Feb 5;11(2):e041427. doi: 10.1136/bmjopen-2020-041427. PMID 33550242